CLINICAL TRIAL: NCT04502043
Title: The Effect of Patients' Characteristics on the Responsiveness to Exercise Therapy for the Management of Femoroacetabular Impingement Syndrome: a Multi-center, Single-group, Intervention Study
Brief Title: Exercise Therapy for Femoroacetabular Impingement Syndrome
Acronym: SWEaT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Schulthess Klinik (Other)
Collaborators: Kantonsspital Winterthur KSW (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SchulthessKlinik
Record Dates: First submitted 2019-06-14; First posted 2020-08-06 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Femoroacetabular Impingement Syndrome
MeSH Terms: conditions — Femoracetabular Impingement | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise therapy (Experimental): Exercise therapy consists of improving dynamic hip joint stability by means of hip-specific and functional lower limb strengthening, core stability and postural balance exercises.
  Interventions: Other: Exercise therapy

INTERVENTIONS:
Other: Exercise therapy — * Education
  * Hip-specific strengthening exercises
  * Functional lower limb strengthening exercises
  * Core stability exercises
  * Postural balance exercises

SUMMARY:
The aim of the clinical trial is to investigate the characteristics of patients, who respond vs. not respond to exercise therapy for the nonsurgical management of femoroacetabular impingement syndrome (FAIS).

DETAILED DESCRIPTION:
Patients with a diagnosis of FAIS will be recruited from 2 clinical centers and will receive exercise therapy (study intervention). Exercise therapy is a semi-standardized intervention and will last 12 weeks (3 months). Hip pain, function and quality of life will be assessed using a patient-reported questionnaire at baseline, 3, 6 and 12 months' follow-up. Hip joint contact pressure will be evaluated using motion analysis and modelling at baseline, 3 and 12 months' follow-up. Hip morphology will be evaluated using imaging at baseline and hip surgery rate will be evaluated at 6 and 12 months' follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 50 years;
* Diagnosis of FAIS;
* Availability of magnetic resonance arthrography and anteroposterior pelvic radiography of the involved hip;
* Signed informed consent form.

Exclusion Criteria:

* Previous hip surgery;
* Any surgery on the lower extremities in the last 6 months;
* Hip dysplasia: lateral center edge angle <25°;
* Hip osteoarthritis: Tönnis grade >1;
* BMI: >35 kg/m2;
* Significant cardiopulmonary diseases.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Change in hip pain, function and quality of life | Baseline to 6 months' follow-up
  Hip pain, function and quality of life will be assessed using the International Hip Outcome Tool - 33 Items

SECONDARY OUTCOMES:
Change in hip pain, function and quality of life | Baseline to 12 months' follow-up
  Hip pain, function and quality of life will be assessed using the International Hip Outcome Tool - 33 Items
Change in hip pain, function and quality of life | Baseline to 3 months' follow-up
  Hip pain, function and quality of life will be assessed using the International Hip Outcome Tool - 33 Items
Change in hip joint contact stress | Baseline to 3 months' follow-up
  Hip joint contact pressure will be assessed using modelling
Change in hip joint contact stress | Baseline to 12 months' follow-up
  Hip joint contact pressure will be assessed using modelling
Hip morphology | Baseline
  Hip morphology will be assessed using imaging
Change in sport activity level | Baseline to 3 months' follow-up
  Sport activity level will be assessed using the Hip Sports Activity Scale
Change in sport activity level | Baseline to 6 months' follow-up
  Sport activity level will be assessed using the Hip Sports Activity Scale
Change in sport activity level | Baseline to 12 months' follow-up
  Sport activity level will be assessed using the Hip Sports Activity Scale
Hip surgery rate | 6 months' follow-up
  Number of patients who will decide to undergo hip surgery
Hip surgery rate | 12 months' follow-up
  Number of patients who will decide to undergo hip surgery
Dropout | 3 months' follow-up
  Number of patients who will not complete the non-surgical intervention protocol

CONTACTS AND LOCATIONS:
Overall Officials: Nicola C Casartelli, PhD, Principal Investigator — Schulthess Klinik
Locations (1):
- Schulthess Clinic, Zurich, Switzerland